CLINICAL TRIAL: NCT03936439
Title: Evolution of Ischemic Stroke Subtypes in Hong Kong
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. IP Yiu Ming Bonaventure, Clinical Tutor, Chinese University of Hong Kong
Other Study IDs: crec 2018.645
Record Dates: First submitted 2019-04-24; First posted 2019-05-03 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Stroke; Stroke, Acute; Neurologic Symptoms
Keywords: stroke
MeSH Terms: conditions — Stroke; Neurologic Manifestations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Consecutive stroke patient: All consecutive stroke patients from five time points, i.e. 2004, 2006, 2008, 2010, 2012, 2014, 2016, 2018 are selected for analysis.

SUMMARY:
Stroke is the 4th leading cause of mortality in Hong Kong. It also carries considerable socioeconomical consequences due to disability.

Ischemic stroke can be classified by the TOAST classification, which includes large artery atherosclerosis, cardioembolism, small-artery occlusion and other causes (1). Among which, intracranial atherosclerosis (ICAS) had been major cause of acute ischemic stroke (AIS) in the Asia Pacific. It was estimated as high as 24.1% of AIS or transient ischemic attacks (TIAs) were attributed to ICAS in China (2). Management of ICAS related strokes has been challenging owing to its high rate of recurrence despite medical therapy. Recent randomized clinical trial suggested that aggressive medical therapy may result in reduction in recurrence compared with historical cohorts (3).

Our group has previously observed a 2.5-fold increase in atrial fibrillation related stroke over a 15-year period (4). The inverstigator also observed a decline in ICAS related AIS as well as its recurrent stroke risk throughout the recent years. Possible mechanisms include better management of metabolic risk factors and aggressive secondary prevention. Other possible reasons are increased atrial fibrillation (AF), small vessel disease (SVD) or other stroke mechanisms.

This study is aim to find the evolution of different stroke subtypes in relation to the characteristics of our stroke population over a 15-year period. This may influence territorial prevention strategy.

DETAILED DESCRIPTION:
Five time points, i.e. 2004, 2006, 2008, 2010, 2012, 2014, 2016, 2018 are selected for analysis. All consecutive stroke patients included in the Prince of Wales Hospital stroke registry will be recruited.

Patients will be stratified according to their stroke subtypes with reference to the TOAST classification (1), which includes large artery disease, cardioembolism, small vessel occlusion, other determined causes, undetermined cause or incomplete investigations.

Stroke etiology is determined by stroke neurologists with reference to the history, physical signs, imaging including carotid duplex, transcranial doppler, computer tomography (CT), CT angiogram, magnetic resonance imaging (MRI), MR angiogram, electrocardiography (ECG) and echocardiography. Interobserver variability for stroke mechanism determination will be evaluated.

Pre-defined demographic data including age, gender, smoking status, vascular risk factors including hyperlipidaemia, hypertension, diabetes, prior stroke or TIA, etc. will be retrieved from the stroke registry.

The investigator will also compare the use of antiplatelet agents, anticoagulants, lipid-lowering agents, specific antihypertensives in the Shatin territory across the 15-year period using the CDARS.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive Chinese stroke patients included in the Prince of Wales Hospital stroke registry at 2-year intervals, i.e. from 2004 to 2018

Exclusion Criteria:

1. Uncertain diagnosis of stroke
2. Non-Chinese patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients in the stroke registry of the Prince of Wales Hospital in the recent 15 years.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Actual)
Dates: Start 2019-03-07 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of ischemic stroke subtype in Hong Kong with the advancement of primary care of cardiovascular control. | 31 Jul, 2019
  Stroke subtypes of the patients in the past 15 years will be classified by the reference of TOAST classification.

SECONDARY OUTCOMES:
The changes of stroke etiology in the population over 15-year period in Hong Kong | 31 Dec, 2019
  Stroke etiology will be determined by the imaging including carotid duplex, transcranial doppler, computer tomography (CT), CT angiogram, magnetic resonance imaging (MRI), MR angiogram, electrocardiography (ECG) and echocardiography.

CONTACTS AND LOCATIONS:
Overall Officials: Yiu Ming Bonaventure IP, MBChB, MRCP, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No